CLINICAL TRIAL: NCT05351515
Title: Prevalence of Non-alcoholic Fatty Liver Disease Among Non-obese Obstructive Sleep Apnea by Using Transient Elastography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Professor, Chinese University of Hong Kong
Other Study IDs: OSA-fattyliver2
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Sleep Apnea, Obstructive; Fatty Liver
MeSH Terms: conditions — Sleep Apnea, Obstructive; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obstructive sleep apnea (OSA) and non-alcoholic fatty liver disease (NAFLD) are both common diseases related to metabolic diseases with potential cardiovascular consequences and liver complications respectively. Though studies show OSA may take part in the progression of hepatic steatosis, the independent contribution of OSA on liver fat accumulation is unknown. It is hypothesized that nocturnal intermittent hypoxia from OSA is the main driver of NAFLD in non-obese OSA patients. This study is to assess the effect of OSA on NAFLD in non-obese patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or more

Exclusion Criteria:

* underlying cause of liver disease
* history of excessive alcoholic consumption (more than 30 g/day for men and 20 g/day for women)
* secondary causes of hepatic steatosis (such as chronic use of systemic corticosteroids)
* positive hepatitis B surface antigen, anti-hepatitis C virus antibody, or histological evidence of other concomitant chronic liver diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is proposed to recruit consecutive patients who have been referred to the Respiratory Clinic at the Prince of Wales Hospital with clinical suspicion of sleep-disordered breathing. In order to invite subjects without symptoms of sleep apnea, collaboration with the Jockey Club School of Public Health and Primary Care, CUHK, to engage healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects found to have fatty liver disease among obese patients with obstructive sleep apnea | baseline
Number of subjects found to have fatty liver disease among non-obese patients with obstructive sleep apnea | baseline

SECONDARY OUTCOMES:
Number of subjects found to have fatty liver disease among obese subjects without obstructive sleep apnea | baseline
Number of subjects found to have fatty liver disease among non-obese subjects without obstructive sleep apnea | baseline
mesenteric fat thickness by ultrasound scan of all subjects | baseline

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, Study Chair — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No